CLINICAL TRIAL: NCT05970978
Title: A Multicenter, Open-label Study to Evaluate the Efficacy and Safety of IBI112 in Participants With Psoriasis Who Were Treated With Biologics and Switched to IBI112
Brief Title: A Study of IBI112 in Chinese Patients With Psoriasis Who Were Previously Treated With Biologics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI112A202CN
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Response to previous biologic therapy (Experimental): Participants with sPGA0 or 1 score and the body surface area affected with psoriasis lesions <3% at baseline; or PASI-75 was achieved after treated with the previous biologics. 200mg of IBI112 will be administered subcutaneously at week 0, 12, 24 and 36.
  Interventions: Drug: regular treatment
- Poor response to previous biologic therapy (Experimental): Participants with sPGA score ≥2 at baseline, or body surface area affected with psoriasis lesions ≥3% at baseline, o PASI-75 was not reached after treated with previous biologics. 200mg of IBI112 will be administered subcutaneously at week 0, 4, 8, 20 and 32.
  Interventions: Drug: Intensive treatment

INTERVENTIONS:
Drug: regular treatment — IBI112 200mg s.c. at week 0, 12, 24 and 36.
  Other Names: Response to previous biologic therapy
  Arms: Response to previous biologic therapy
Drug: Intensive treatment — IBI112 200mg s.c. at week 0, 4, 8, 20 and 32.
  Other Names: Poor response to previous biologic therapy
  Arms: Poor response to previous biologic therapy

SUMMARY:
This is a multicenter, open-label study aim to evaluate the efficacy and safety of IBI112 in Chinese participants with plaque psoriasis who were treated with biologics and switched to IBI112. The study will enroll 160 participants who were diagnosed with plaque psoriasis. The whole study consists of 4 weeks of screening, 32 or 36 weeks of treatment and a safety follow-up visit at Week 44.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old;
2. Evaluated suitable for continuing biologic therapy for plaque psoriasis by the investigator;
3. Received previous biologic therapy with at least 4 months.

Exclusion Criteria:

1. Diagnosed with guttate psoriasis, pustular psoriasis, erythrodermic psoriasis, or drug-induced psoriasis (e.g., psoriasis caused by beta blockers, calcium channel inhibitors, etc.) at screening;
2. Previously treated with IBI112 or other IL-23 inhibitors;
3. Treated with two biologics for psoriasis within 4 months prior to screening;
4. Treated with topical therapy for psoriasis within 2 weeks prior to the first dose administration, or treated with systemic non-biological agents or phototherapy within 4 weeks prior to the first dose administration;
5. Treated with Natalizumab, or B/T cell regulators (e.g., Rituximab, Abatacept, or Visilizumab) within 12 months prior to the first dose administration;
6. Not willing to avoid constant sunshine and other ultraviolet light sources exposure during the study;
7. Treated with an investigational biologic within 6 months prior to the first dose administration, or any investigational therapy within 30 days, or an investigational drug within 5 half-lives, or currently participating in a clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who achieve sPGA clean (0) or nearly clean (1) ，and BSA < 3% | Week 16

SECONDARY OUTCOMES:
Percentage of participants who achieve sPGA clean (0) at Week 16. | Week 16
Percentage of participants with a DLQI score of 0/1 at Week 16. | Week 16
Percentage of participants with sPGA 0/1 or sPGA 0 or DLQI 0/1 at Week 44. | Week 44
Percentage of participants who achieve sPGA 0 or 1 at week 16 and maintain that up to Week 44 | Week 16 up to Week 44

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital of Shandong First Medical University (Shandong Provincial Hospitial of Dermatology), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Q, Yang B, Gu H, Wu L, Qin L, Wang L, Li Y, Gu L, Shen Z, Zhang S, Lu J, Shi Y, Tao X, Cui Y, Zhang S, Ren H, Li L, Man X, Chen H, Xiao R, Yang Z, Ren Y, Ye R, Du H, Zhang F. Efficacy and Safety of Switching to Picankibart from Non-interleukin-23 Subunit p19 Inhibitors in Patients with Plaque Psoriasis: A Multicenter, Open-Label, Phase 2 Trial. Adv Ther. 2026 Jan 27. doi: 10.1007/s12325-025-03419-w. Online ahead of print. PMID 41591649